CLINICAL TRIAL: NCT04675957
Title: Cardiac Rehab Retrospective Review (CR3)
Acronym: CR3
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0204
Record Dates: First submitted 2020-10-19; First posted 2020-12-19 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Sudden Cardiac Death; Heart Failure; Ventricular Arrythmia; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: wearable cardioverter-defibrillator; cardiac rehabilitation
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Failure; Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cardiac rehabilitation — stationary or ambulatory cardiac rehabilitation

SUMMARY:
All patients enrolled in the Austrian LifeVest Registry will be retrospectively screened for successfully completed ambulatory or stationary rehabilitation program. Baseline characteristics, complete rehab data, outcomes and follow up data, as well as wearable cardioverter defibrillator(WCD)-derived data will be collected from these patients.

Specifically, performance data from the start of the exercise training (ET) will be compared to the end of ET; including type of training, exertion, time and duration will be collected. In addition, WCD recorded data such as automatically and manually recorded ECGs, compliance, and TRENDS data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed WCD as part of the Austrian WCD registry population from 2014-2018
* Partial (>50%) or full completion of a rehabilitation program when wearing the WCD in Austria
* ≥18 years old and able to give informed consent

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Austrian patients with a WCD having the TRENDS feature who underwent cardiac rehabilitation from 2014-18 will be retrospectively analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Number of Arrhythmias (as recorded by clinic or WCD) | 3 months
  To investigate the safety and feasibility of WCD therapy during cardiac rehabilitation, the following data on Arrhythmias captured via WCD or Surface ECG will be collected:
  * Atrial tachycardia
  * Ventricular tachycardia
  * Bradycardia
Number of adequate WCD alarms (as recorded by WCD) per patient | 3 months
  To investigate the safety and feasibility of WCD therapy during cardiac rehabilitation, the number of adequate WCD alarms will be recorded
Number of inadequate WCD alarms (as recorded by WCD) per patient | 3 months
  To investigate the safety and feasibility of WCD therapy during cardiac rehabilitation, the number of inadequate WCD alarms will be recorded
Number of patients with appropriate WCD Shocks | 3 months
  To investigate the safety and feasibility of WCD therapy during cardiac rehabilitation, the number of appropriate WCD shocks will be collected.
Number of patients with Syncopes/Presyncopes | 3 months
  To investigate the safety and feasibility of WCD therapy during cardiac rehabilitation, data of Syncopes or Pre-Syncopes will be collected.
Number of patients with abnormal blood pressure (measured in mmHg) | 3 months
  To investigate the safety and feasibility of WCD therapy during cardiac rehabilitation, the following data for abnormal blood pressure will be collected:
  * Occurrence of Hypotension
  * Occurrence of Hypertension
Number of other issues with WCD | 3 months
  To investigate the safety and feasibility of WCD therapy during cardiac rehabilitation, every data with an issue with WCD disturbing the normal rehabilitation activities will be collected.
Number of other Adverse Events | 3 months
  To investigate the safety and feasibility of WCD therapy during cardiac rehabilitation, other adverse events recorded by staff during therapy session that stopped ET session (notWCD specific) will be collected.
Number of patients with inappropriate WCD Shocks | 3 months
  To investigate the safety and feasibility of WCD therapy during cardiac rehabilitation, the number of inappropriate WCD shocks (captured via LifeVestNetwork) will be collected.

SECONDARY OUTCOMES:
Difference in physical exercise capacity - measured in METs | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
Performance in ergometry - measured in watts (difference between initial Evaluation and final Evaluation) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
Body weight - measured in kilogram (difference between initial Evaluation and final Evaluation) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
Body Mass Index (BMI, weight and height will be combined to report BMI in kg/m^2); (difference between initial Evaluation and final Evaluation) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
Blood pressure - measured in mmHg (difference between initial Evaluation and final Evaluation) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
Left ventricular ejection fraction - measured in % (difference between initial Evaluation and final Evaluation) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
  With echocardiography the left ventricular ejection fraction (%) will be collected.
Left ventricular end diastolic diameter (measured in mm) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
  With Echocardiography Left ventricular end diastolic diameter (mm) will be collected.
Size of the Left atrial (measured in mm) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
  With Echocardiography. the size of the Left atrial (mm) will be collected.
Right atrial diameter (measured in mm) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
  With Echocardiography, Right atrial diameter (mm) will be collected.
diastolic dysfunction (measured in grade) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
  With Echocardiography, the diastolic dysfunction (grade) will be collected.
Intraventricular septum (diastolic, measured in mm) | 3 months
  The measures regarding exercise performance while wearing a WCD during cardiac rehabilitation will be evaluated through the use of descriptive statistics before and after rehabilitation.
  With Echocardiography, the Intraventricular septum (diastole, mm) will be collected.
Heart rate derived from the WCD (measured in beats per Minute) | 3 months
  The correlation of WCD-derived parameters such as heart rate with patients' exercise performance during cardiac rehabilitation will primarily be an ad-hoc statistical analyses.
Body Position derived from the WCD | 3 months
  The correlation of WCD-derived parameters such as body position with patients' exercise performance during cardiac rehabilitation will primarily be an ad-hoc statistical analyses. Body position is measured by position sensors.
Step count derived from the WCD (steps/day) | 3 months
  The correlation of WCD-derived parameters such as the step count with patients' exercise performance during cardiac rehabilitation will primarily be an ad-hoc statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Scherr, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rohrer U, Reischl A, Manninger M, Binder RK, Fiedler L, Gruska M, Altenberger J, Dorr A, Steinwender C, Stuehlinger M, Wonisch M, Zirngast B, Zweiker D, Zirlik A, Scherr D; Austrian WCD Study Group. Cardiovascular Rehabilitation With a WCD-Data From the CR3 Study (Cardiac Rehab Retrospective Review). J Cardiopulm Rehabil Prev. 2024 Mar 1;44(2):115-120. doi: 10.1097/HCR.0000000000000832. Epub 2023 Nov 30. PMID 38032261